CLINICAL TRIAL: NCT01401166
Title: A Randomized, Multi-Center Cross-Over Study to Evaluate Patient Preference and Health Care Professional (HCP) Satisfaction With Subcutaneous (SC) Administration of Trastuzumab in HER2-Positive Early Breast Cancer (EBC)
Brief Title: Participant Preference of Subcutaneous (SC) Versus Intravenous (IV) Herceptin (Trastuzumab) in Human Epidermal Growth Factor Receptor (HER) 2-Positive Early Breast Cancer
Acronym: PrefHER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: MO22982; 2010-024099-25 (EudraCT Number)
Record Dates: First submitted 2011-07-22; First posted 2011-07-25 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

ARMS (4):
- Cohort 1: SC (SID) then IV Herceptin (Experimental): Participants will receive Herceptin on Day 1 of each 3-week cycle for 18 cycles. During Cycles 1 to 4 of the crossover period, SC Herceptin will be administered via single-use injection device (SID), and during Cycles 5 to 8, IV Herceptin will be given. In the continuation period, participants will receive IV Herceptin for up to 10 remaining cycles. Administration will be performed by HCP. Those with at least 2 treatment cycles remaining of the 18-cycle treatment course after the crossover period will be offered the opportunity to self-administer SC Herceptin via SID under the direction of a trained HCP.
  Interventions: Drug: Herceptin; Device: Single-Use Injection Device
- Cohort 1: IV then SC (SID) Herceptin (Experimental): Participants will receive Herceptin on Day 1 of each 3-week cycle for 18 cycles. During Cycles 1 to 4 of the crossover period, IV Herceptin will be given, and during Cycles 5 to 8, SC Herceptin will be administered via SID. In the continuation period, participants will receive IV Herceptin for up to 10 remaining cycles. Administration will be performed by HCP. Those with at least 2 treatment cycles remaining of the 18-cycle treatment course after the crossover period will be offered the opportunity to self-administer SC Herceptin via SID under the direction of a trained HCP.
  Interventions: Drug: Herceptin; Device: Single-Use Injection Device
- Cohort 2: SC (Vial) then IV Herceptin (Experimental): Participants will receive Herceptin on Day 1 of each 3-week cycle for 18 cycles. During Cycles 1 to 4 of the crossover period, SC Herceptin will be administered via handheld syringe using the vial formulation, and during Cycles 5 to 8, IV Herceptin will be given. In the continuation period, participants will receive SC Herceptin via handheld syringe using the vial formulation for up to 10 remaining cycles. Administration will be performed by HCP throughout the study.
  Interventions: Drug: Herceptin
- Cohort 2: IV then SC (Vial) Herceptin (Experimental): Participants will receive Herceptin on Day 1 of each 3-week cycle for 18 cycles. During Cycles 1 to 4 of the crossover period, IV Herceptin will be given, and during Cycles 5 to 8, SC Herceptin will be administered via handheld syringe using the vial formulation. In the continuation period, participants will receive SC Herceptin via handheld syringe using the vial formulation for up to 10 remaining cycles. Administration will be performed by HCP throughout the study.
  Interventions: Drug: Herceptin

INTERVENTIONS:
Drug: Herceptin — Herceptin will be given on Day 1 of each 3-week cycle for a total of 18 cycles. If study treatment for Cycle 1 is IV Herceptin, the initial dose will be a loading dose of 8 milligrams per kilogram (mg/kg) for de novo participants who start Herceptin treatment in the study. For all other cycles where IV Herceptin is given and for non-de novo participants, the dose will be 6 mg/kg. The SC dose will be 600 milligrams (mg) for both the SID and vial formulations for all cycles where SC Herceptin is given.
  Other Names: Trastuzumab
  Arms: Cohort 1: SC (SID) then IV Herceptin
Drug: Herceptin — Herceptin will be given on Day 1 of each 3-week cycle for a total of 18 cycles. If study treatment for Cycle 1 is IV Herceptin, the initial dose will be a loading dose of 8 mg/kg for de novo participants who start Herceptin treatment in the study. For all other cycles where IV Herceptin is given and for non-de novo participants, the dose will be 6 mg/kg. The SC dose will be 600 mg for both the SID and vial formulations for all cycles where SC Herceptin is given.
  Other Names: Trastuzumab
  Arms: Cohort 1: IV then SC (SID) Herceptin; Cohort 2: IV then SC (Vial) Herceptin; Cohort 2: SC (Vial) then IV Herceptin
Device: Single-Use Injection Device — The SID will be used, containing Herceptin 600 mg per 5 milliliters (mL).
  Arms: Cohort 1: SC (SID) then IV Herceptin
Device: Single-Use Injection Device — The SID will be used, containing Herceptin 600 mg per 5 mL.
  Arms: Cohort 1: IV then SC (SID) Herceptin

SUMMARY:
This randomized, open-label, crossover study will evaluate participants' preference and healthcare professional (HCP) satisfaction with SC versus IV Herceptin administration in HER2-positive early breast cancer. Participants will be randomized to receive either SC Herceptin or IV Herceptin every 3 weeks for Cycles 1 to 4, followed by crossover to the other treatment administration for Cycles 5 to 8. For up to 10 additional cycles (for a total of 18 cycles), participants will receive IV or SC Herceptin every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HER2-positive primary breast cancer
* No evidence of residual, locally recurrent, or metastatic disease after completion of surgery and chemotherapy (neo-adjuvant or adjuvant)
* Completed neo-adjuvant chemotherapy prior to entry, if received
* At least 8 remaining cycles out of the total 18 planned 3-week cycles, if received IV Herceptin
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

* History of other malignancy, except for ductal carcinoma in situ of the breast, curatively treated carcinoma in situ of the cervix, basal cell carcinoma, or other curatively treated malignancies of which the participant has been disease-free for at least 5 years
* Inadequate bone marrow function
* Impaired liver function
* Inadequate renal function
* Serious cardiovascular disease
* Human immunodeficiency virus or hepatitis B or C infection
* Prior maximum cumulative dose of doxorubicin greater than (>) 360 milligrams per meter-squared (mg/m^2) or epirubicin >720 mg/m^2 or equivalent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (71):
- Canada (6):
  - Barrie, Ontario
  - Brampton, Ontario
  - Kitchener, Ontario
  - Sault Ste. Marie, Ontario
  - Toronto, Ontario
  - Saskatoon, Saskatchewan
- Denmark (3):
  - Herning
  - Odense
  - Vejle
- France (11):
  - Besançon
  - Bobigny
  - Bordeaux
  - Caen
  - La Tronche
  - LeMans
  - Lyon
  - Paris
  - Rennes
  - Saint-Cloud
  - Strasbourg
- Germany (11):
  - Berlin
  - Deggendorf
  - Essen
  - Fürstenwalde
  - Hamburg
  - Hanover
  - Magedburg
  - Mainz
  - Meiningen
  - Recklinghausen
  - Ulm
- Italy (5):
  - Genoa, Liguria
  - Milan, Lombardy
  - Pavia, Lombardy
  - Antella (FI), Tuscany
  - Terni, Umbria
- Poland (2):
  - Gdansk
  - Warsaw
- Russia (6):
  - Irkutsk
  - Kazan'
  - Moscow
  - Orenburg
  - Saint Petersburg
  - Yekaterinburg
- Spain (10):
  - Barcelona, Barcelona
  - Córdoba, Cordoba
  - Guadalajara, Guadalajara
  - Huesca, Huesca
  - Madrid, Madrid
  - Málaga, Malaga
  - Oviedo, Principality of Asturias
  - Seville, Sevilla
  - Barakaldo, Vizcaya
  - Zamora, Zamora
- Sweden (4):
  - Eskilstuna
  - Gävle
  - Jönköping
  - Sundsvall
- Switzerland (2):
  - Baden
  - Zurich
- Turkey (Türkiye) (4):
  - Adana
  - Ankara
  - Bornova, ?zm?r
  - Gaziantep
- United Kingdom (7):
  - Brighton
  - Cardiff
  - Chelmsford
  - Maidstone
  - Nottingham
  - Peterborough
  - Truro

REFERENCES:
- [Derived] Pivot X, Verma S, Fallowfield L, Muller V, Lichinitser M, Jenkins V, Sanchez Munoz A, Machackova Z, Osborne S, Gligorov J; PrefHer Study Group. Efficacy and safety of subcutaneous trastuzumab and intravenous trastuzumab as part of adjuvant therapy for HER2-positive early breast cancer: Final analysis of the randomised, two-cohort PrefHer study. Eur J Cancer. 2017 Nov;86:82-90. doi: 10.1016/j.ejca.2017.08.019. Epub 2017 Sep 28. PMID 28963915
- [Derived] Gligorov J, Curigliano G, Muller V, Knoop A, Jenkins V, Verma S, Osborne S, Lauer S, Machackova Z, Fallowfield L, Pivot X. Switching between intravenous and subcutaneous trastuzumab: Safety results from the PrefHer trial. Breast. 2017 Aug;34:89-95. doi: 10.1016/j.breast.2017.05.004. Epub 2017 May 23. PMID 28549309
- [Derived] De Cock E, Pivot X, Hauser N, Verma S, Kritikou P, Millar D, Knoop A. A time and motion study of subcutaneous versus intravenous trastuzumab in patients with HER2-positive early breast cancer. Cancer Med. 2016 Mar;5(3):389-97. doi: 10.1002/cam4.573. Epub 2016 Jan 25. PMID 26806010
- [Derived] Pivot X, Gligorov J, Muller V, Curigliano G, Knoop A, Verma S, Jenkins V, Scotto N, Osborne S, Fallowfield L; PrefHer Study Group. Patients' preferences for subcutaneous trastuzumab versus conventional intravenous infusion for the adjuvant treatment of HER2-positive early breast cancer: final analysis of 488 patients in the international, randomized, two-cohort PrefHer study. Ann Oncol. 2014 Oct;25(10):1979-1987. doi: 10.1093/annonc/mdu364. Epub 2014 Jul 28. PMID 25070545
- [Derived] Pivot X, Gligorov J, Muller V, Barrett-Lee P, Verma S, Knoop A, Curigliano G, Semiglazov V, Lopez-Vivanco G, Jenkins V, Scotto N, Osborne S, Fallowfield L; PrefHer Study Group. Preference for subcutaneous or intravenous administration of trastuzumab in patients with HER2-positive early breast cancer (PrefHer): an open-label randomised study. Lancet Oncol. 2013 Sep;14(10):962-70. doi: 10.1016/S1470-2045(13)70383-8. Epub 2013 Aug 19. PMID 23965225

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 248 participants were randomized into the study in Cohort 1 (of whom 244 were treated) and 240 participants were randomized into the study in Cohort 2 (of whom 239 were treated). Those participants who did not receive any treatment were not included in the treatment periods of the Participant Flow.
Groups:
- Cohort 1: SC (SID) Then IV Herceptin: Participants received Herceptin on Day 1 of each 3-week cycle for 18 cycles. During Cycles 1 to 4 of the crossover period, SC Herceptin was administered via single-use injection device (SID), and during Cycles 5 to 8, IV Herceptin was given. In the continuation period, participants received IV Herceptin for up to 10 remaining cycles. Administration was performed by healthcare professional (HCP). Those with at least 2 treatment cycles remaining of the 18-cycle treatment course after the crossover period were offered the opportunity to self-administer SC Herceptin via SID under the direction of a trained HCP. The SC dose was 600 milligrams (mg) for all cycles where SC Herceptin was given, and the IV dose was 6 milligrams per kilogram (mg/kg) for all cycles where IV Herceptin was given.
- Cohort 1: IV Then SC (SID) Herceptin: Participants received Herceptin on Day 1 of each 3-week cycle for 18 cycles. During Cycles 1 to 4 of the crossover period, IV Herceptin was given, and during Cycles 5 to 8, SC Herceptin was administered via SID. In the continuation period, participants received IV Herceptin for up to 10 remaining cycles. Administration was performed by HCP. Those with at least 2 treatment cycles remaining of the 18-cycle treatment course after the crossover period were offered the opportunity to self-administer SC Herceptin via SID under the direction of a trained HCP. The IV dose was a loading dose of 8 mg/kg in Cycle 1 for de novo participants who started Herceptin treatment in the study, and a dose of 6 mg/kg for all subsequent cycles where IV Herceptin was given and for non-de novo participants. The SC dose was 600 mg for all cycles where SC Herceptin was given.
- Cohort 2: SC (Vial) Then IV Herceptin: Participants received Herceptin on Day 1 of each 3-week cycle for 18 cycles. During Cycles 1 to 4 of the crossover period, SC Herceptin was administered via handheld syringe using the vial formulation, and during Cycles 5 to 8, IV Herceptin was given. In the continuation period, participants received SC Herceptin via handheld syringe using the vial formulation for up to 10 remaining cycles. Administration was performed by HCP throughout the study. The SC dose was 600 mg for all cycles where SC Herceptin was given, and the IV dose was 6 mg/kg for all cycles where IV Herceptin was given.
- Cohort 2: IV Then SC (Vial) Herceptin: Participants received Herceptin on Day 1 of each 3-week cycle for 18 cycles. During Cycles 1 to 4 of the crossover period, IV Herceptin was given, and during Cycles 5 to 8, SC Herceptin was administered via handheld syringe using the vial formulation. In the continuation period, participants received SC Herceptin via handheld syringe using the vial formulation for up to 10 remaining cycles. Administration was performed by HCP throughout the study. The IV dose was a loading dose of 8 mg/kg in Cycle 1 for de novo participants who started Herceptin treatment in the study, and a dose of 6 mg/kg for all subsequent cycles where IV Herceptin was given and for non-de novo participants. The SC dose was 600 mg for all cycles where SC Herceptin was given.
Period: Crossover Treatment 1 (Cycles 1 to 4)
Arm/Group | Cohort 1: SC (SID) Then IV Herceptin | Cohort 1: IV Then SC (SID) Herceptin | Cohort 2: SC (Vial) Then IV Herceptin | Cohort 2: IV Then SC (Vial) Herceptin
Started | 122 (A total of 124 participants were randomized, but 2 did not receive any treatment.) | 122 (A total of 124 participants were randomized, but 2 did not receive any treatment.) | 121 (A total of 121 participants were randomized who all received study treatment.) | 118 (A total of 119 participants were randomized, but 1 did not receive any treatment.)
Completed | 119 | 120 | 119 | 116
Not Completed | 3 | 2 | 2 | 2
Period: Crossover Treatment 2 (Cycles 5 to 8)
Arm/Group | Cohort 1: SC (SID) Then IV Herceptin | Cohort 1: IV Then SC (SID) Herceptin | Cohort 2: SC (Vial) Then IV Herceptin | Cohort 2: IV Then SC (Vial) Herceptin
Started | 119 | 120 | 119 | 116
Completed | 113 | 116 | 107 | 105
Not Completed | 6 | 4 | 12 | 11
Period: Continuation Treatment (Cycles 9 to 18)
Arm/Group | Cohort 1: SC (SID) Then IV Herceptin | Cohort 1: IV Then SC (SID) Herceptin | Cohort 2: SC (Vial) Then IV Herceptin | Cohort 2: IV Then SC (Vial) Herceptin
Started | 113 | 116 | 107 | 105
Completed | 109 | 109 | 105 | 102
Not Completed | 4 | 7 | 2 | 3
Period: Safety Follow-Up Period
Arm/Group | Cohort 1: SC (SID) Then IV Herceptin | Cohort 1: IV Then SC (SID) Herceptin | Cohort 2: SC (Vial) Then IV Herceptin | Cohort 2: IV Then SC (Vial) Herceptin
Started | 124 (All 124 randomized participants entered follow-up regardless of whether they received treatment.) | 124 (All 124 randomized participants entered follow-up regardless of whether they received treatment.) | 121 (All 121 randomized participants entered follow-up regardless of whether they received treatment.) | 119 (All 119 randomized participants entered follow-up regardless of whether they received treatment.)
Completed | 99 | 106 | 104 | 100
Not Completed | 25 | 18 | 17 | 19

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who received at least one dose of Herceptin.
Groups:
- Cohort 1 Overall: SC (SID) and IV Herceptin: Participants received Herceptin on Day 1 of each 3-week cycle for 18 cycles, randomized to one of two crossover sequences: SC Herceptin via SID for Cycles 1 to 4 followed by IV Herceptin for Cycles 5 to 8, or vice versa. In the continuation period, participants received IV Herceptin for up to 10 remaining cycles. Administration was performed by HCP. Those with at least 2 treatment cycles remaining of the 18-cycle treatment course after the crossover period were offered the opportunity to self-administer SC Herceptin via SID under the direction of a trained HCP. If study treatment for Cycle 1 was IV Herceptin, the initial dose was a loading dose of 8 mg/kg for de novo participants who started Herceptin treatment in the study. For all other cycles where IV Herceptin was given and for non-de novo participants, the dose was 6 mg/kg. The SC dose was 600 mg for all cycles where SC Herceptin was given.
- Cohort 2 Overall: SC (Vial) and IV Herceptin: Participants received Herceptin on Day 1 of each 3-week cycle for 18 cycles, randomized to one of two crossover sequences: SC Herceptin via handheld syringe using the vial formulation for Cycles 1 to 4 followed by IV Herceptin for Cycles 5 to 8, or vice versa. In the continuation period, participants received SC Herceptin for up to 10 remaining cycles. Administration was performed by HCP throughout the study. If study treatment for Cycle 1 was IV Herceptin, the initial dose was a loading dose of 8 mg/kg for de novo participants who started Herceptin treatment in the study. For all other cycles where IV Herceptin was given and for non-de novo participants, the dose was 6 mg/kg. The SC dose was 600 mg for all cycles where SC Herceptin was given.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Overall: SC (SID) and IV Herceptin | Cohort 2 Overall: SC (Vial) and IV Herceptin | Total
Number analyzed (Participants) | 244 | 239 | 483
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (11.40) | 52.9 (10.87) | 53.1 (11.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 244 | 239 | 483
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants by Preferred Method of Drug Administration
Description: The preferred method of drug administration (IV or SC Herceptin) was assessed in trial-specific telephone interviews with each study participant. Participants were asked, "All things considered, which method of administration did you prefer?" at the end of the crossover period (Week 24). The percentage of participants who preferred each method of drug administration was reported.
Time Frame: Week 24
Population: Intent-to-Treat (ITT) Population: All participants who received both IV and SC Herceptin and who completed the trial-specific telephone interview conducted after the end of the crossover period.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 1: SC (SID) Then IV Herceptin: Participants received Herceptin on Day 1 of each 3-week cycle for 18 cycles. During Cycles 1 to 4 of the crossover period, SC Herceptin was administered via SID, and during Cycles 5 to 8, IV Herceptin was given. In the continuation period, participants received IV Herceptin for up to 10 remaining cycles. Administration was performed by HCP. Those with at least 2 treatment cycles remaining of the 18-cycle treatment course after the crossover period were offered the opportunity to self-administer SC Herceptin via SID under the direction of a trained HCP. The SC dose was 600 mg for all cycles where SC Herceptin was given, and the IV dose was 6 mg/kg for all cycles where IV Herceptin was given.
Arm/Group | Cohort 1: SC (SID) Then IV Herceptin | Cohort 1: IV Then SC (SID) Herceptin | Cohort 2: SC (Vial) Then IV Herceptin | Cohort 2: IV Then SC (Vial) Herceptin
Number analyzed (Participants) | 117 | 119 | 118 | 113
percentage of participants
  SC Herceptin | 95.7 | 87.4 | 83.9 | 88.5
  IV Herceptin | 4.3 | 9.2 | 13.6 | 11.5
  No Preference | 0.0 | 3.4 | 2.5 | 0.0
Statistical Analysis 1: Comparison: Cohort 1: SC (SID) Then IV Herceptin; Test type: Superiority or Other; Estimated Proportion = 0.957, 95% CI 2-sided [0.903 to 0.986] — The estimated proportion of participants who preferred SC Herceptin and the corresponding exact binomial confidence interval (CI) were determined
Statistical Analysis 2: Comparison: Cohort 1: SC (SID) Then IV Herceptin; Test type: Superiority or Other; Estimated Proportion = 0.964, 95% CI 2-sided [0.908 to 0.986] — The estimated proportion of participants who preferred SC Herceptin and the corresponding CI were determined using logistic regression with factors of previous Herceptin status and treatment
Statistical Analysis 3: Comparison: Cohort 1: IV Then SC (SID) Herceptin; Test type: Superiority or Other; Estimated Proportion = 0.874, 95% CI 2-sided [0.801 to 0.928] — The estimated proportion of participants who preferred SC Herceptin and the corresponding exact binomial CI were determined
Statistical Analysis 4: Comparison: Cohort 1: IV Then SC (SID) Herceptin; Test type: Superiority or Other; Estimated Proportion = 0.892, 95% CI 2-sided [0.804 to 0.943] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Cohort 2: SC (Vial) Then IV Herceptin; Test type: Superiority or Other; Estimated Proportion = 0.839, 95% CI 2-sided [0.760 to 0.900] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 6: Comparison: Cohort 2: SC (Vial) Then IV Herceptin; Test type: Superiority or Other; Estimated Proportion = 0.874, 95% CI 2-sided [0.776 to 0.933] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Cohort 2: IV Then SC (Vial) Herceptin; Test type: Superiority or Other; Estimated Proportion = 0.885, 95% CI 2-sided [0.811 to 0.937] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 8: Comparison: Cohort 2: IV Then SC (Vial) Herceptin; Test type: Superiority or Other; Estimated Proportion = 0.911, 95% CI 2-sided [0.827 to 0.956] — [estimate comment as in outcome 1, analysis 2]

2. Secondary Outcome: Percentage of HCPs by Most Satisfied Method of Drug Administration
Description: The method of drug administration with which HCPs were most satisfied (IV or SC Herceptin) was assessed via questionnaire with each HCP using the question, "All things considered, with which method of administration were you most satisfied?" at the end of the crossover period (Week 24). The percentage of HCPs who were most satisfied with each method of drug administration was reported.
Time Frame: Week 24
Population: HCP Population: All HCPs who participated in the study and completed the HCP questionnaire. Results were planned to be analyzed for all HCPs combined because the objective of the study was to compare preference between SC and IV Herceptin.
Measure: Number; unit: percentage of HCPs
Units Other Than Participants: HCPs
Groups:
- All HCPs: SC and IV Herceptin: Participants received Herceptin on Day 1 of each 3-week cycle for 18 cycles, randomized to one of two crossover sequences: SC Herceptin via SID (Cohort 1) or vial (Cohort 2) for Cycles 1 to 4 followed by IV Herceptin for Cycles 5 to 8, or vice versa. In the continuation period, participants received IV Herceptin (Cohort 1) or SC Herceptin (Cohort 2) for up to 10 remaining cycles. Participants in Cohort 1 with at least 2 treatment cycles remaining of the 18-cycle treatment course after the crossover period were offered to self-administer SC Herceptin via SID under the direction of a trained HCP, whereas in Cohort 2, administration was performed by HCP throughout the study. If study treatment for Cycle 1 was IV Herceptin, the initial dose was a loading dose of 8 mg/kg for de novo participants who started Herceptin treatment in the study. For all other cycles where IV Herceptin was given and for non-de novo participants, the dose was 6 mg/kg. The SC dose was 600 mg for both SID and vial.
Arm/Group | All HCPs: SC and IV Herceptin
Number analyzed (Participants) | 235
Number analyzed (HCPs) | 235
percentage of HCPs
  SC Herceptin | 77.0
  IV Herceptin | 3.0
  No Preference | 20.0

3. Secondary Outcome: Percentage of HCPs by Time Required to Perform Each Method of Drug Administration
Description: The time required to perform each method of drug administration was assessed via questionnaire with each HCP by asking to rate the amount of time it took to administer each method of drug administration (IV or SC Herceptin) at the end of the crossover period (Week 24). Time was rated in the following time block categories: less than (<) 5 minutes, 6 to 10 minutes, 11 to 15 minutes, 16 to 20 minutes, and greater than (>) 20 minutes. Responses of "Not Sure" and "Unknown" were also allowed. The percentage of HCPs who rated the amount of time in each of the categories was reported.
Time Frame: Week 24
Population: HCP Population. Results were planned to be analyzed for all HCPs combined because the objective of the study was to compare HCP perceived time savings with use of SC over IV Herceptin.
Measure: Number; unit: percentage of HCPs
Units Other Than Participants: HCPs
Arm/Group | All HCPs: SC and IV Herceptin
Number analyzed (Participants) | 235
Number analyzed (HCPs) | 235
percentage of HCPs
  SC Herceptin, <5 minutes | 44.3
  SC Herceptin, 6 to 10 minutes | 46.4
  SC Herceptin, 11 to 15 minutes | 3.4
  SC Herceptin, 16 to 20 minutes | 0.4
  SC Herceptin, >20 minutes | 0.4
  SC Herceptin, Not Sure | 0.0
  SC Herceptin, Unknown | 5.1
  IV Herceptin, <5 minutes | 11.1
  IV Herceptin, 6 to 10 minutes | 9.8
  IV Herceptin, 11 to 15 minutes | 3.8
  IV Herceptin, 16 to 20 minutes | 44.3
  IV Herceptin, >20 minutes | 22.1
  IV Herceptin, Not Sure | 5.1
  IV Herceptin, Unknown | 3.8

4. Secondary Outcome: Percentage of Participants With an Event-Free Survival (EFS) Event
Description: EFS events included local, regional, or distant recurrence of the original breast cancer, occurrence of contralateral breast cancer, or death due to any cause. The percentage of participants who had an EFS event at any time on study was reported.
Time Frame: From Baseline until time of event; assessed every 6 months (median follow-up of 3 years)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: SC (SID) Then IV Herceptin | Cohort 1: IV Then SC (SID) Herceptin | Cohort 2: SC (Vial) Then IV Herceptin | Cohort 2: IV Then SC (Vial) Herceptin
Number analyzed (Participants) | 117 | 119 | 118 | 113
percentage of participants | 13.7 | 6.7 | 11.9 | 7.1

5. Secondary Outcome: Duration of EFS According to Kaplan-Meier Estimate
Description: EFS was defined as the time from randomization to a local, regional, or distant recurrence of the original breast cancer, occurrence of contralateral breast cancer, or death due to any cause. The median duration of EFS and corresponding 95 percent (%) CI according to Kaplan-Meier estimates were planned to be reported and expressed in months.
Time Frame: From Baseline until time of event; assessed every 6 months (median follow-up of 3 years)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: SC (SID) Then IV Herceptin | Cohort 1: IV Then SC (SID) Herceptin | Cohort 2: SC (Vial) Then IV Herceptin | Cohort 2: IV Then SC (Vial) Herceptin
Number analyzed (Participants) | 117 | 119 | 118 | 113
months | NA [NA to NA] — Median and 95% CI not presented due to insufficient follow-up to allow estimation. | NA [42.0 to NA] — Median and 95% CI not presented due to insufficient follow-up to allow estimation. | NA [NA to NA] — Median and 95% CI not presented due to insufficient follow-up to allow estimation. | NA [NA to NA] — Median and 95% CI not presented due to insufficient follow-up to allow estimation.

6. Secondary Outcome: 3-Year EFS Rate
Description: EFS events included local, regional, or distant recurrence of the original breast cancer, occurrence of contralateral breast cancer, or death due to any cause. The proportion of participants without an EFS event (i.e., the EFS rate) and corresponding 95% CI at 3 years after randomization was reported.
Time Frame: Year 3
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Cohort 1: SC (SID) Then IV Herceptin | Cohort 1: IV Then SC (SID) Herceptin | Cohort 2: SC (Vial) Then IV Herceptin | Cohort 2: IV Then SC (Vial) Herceptin
Number analyzed (Participants) | 117 | 119 | 118 | 113
proportion of participants | 0.849 [0.763 to 0.906] | 0.948 [0.887 to 0.976] | 0.886 [0.811 to 0.932] | 0.937 [0.873 to 0.970]

7. Secondary Outcome: Percentage of Participants With Responses of "Agree" or "Strongly Agree" on the SC SID Satisfaction Questionnaire
Description: Participants who performed self-administration of SC Herceptin via SID were given an evaluation questionnaire during the continuation period (Weeks 25 to 52) after their first self-administration. Participants responded to 5 statements about their comfort with self-injection, the convenience of the SID, their self-confidence using the SID, their satisfaction with the SID, and whether they would consider using the SID again in the future. Each statement used a 5-item rating scale with responses from "Strongly Disagree" to "Strongly Agree". The percentage of participants with a positive response (either "Agree" or "Strongly Agree") to each questionnaire statement was reported.
Time Frame: Immediately following first self-administration of SC Herceptin via SID (once during Weeks 25 to 52)
Population: Safety Population. The "Number of Participants Analyzed" reflects those who self-administered SC Herceptin using the SID and completed the SC SID questionnaire. Results were planned to be analyzed for only Cohort 1 because the objective of the study was to evaluate satisfaction among those who self-administered the SID formulation of Herceptin.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: SC (SID) Then IV Herceptin | Cohort 1: IV Then SC (SID) Herceptin
Number analyzed (Participants) | 19 | 15
percentage of participants
  Comfortable | 94.7 | 86.7
  Convenient | 100 | 100
  Confident | 100 | 100
  Satisfied | 100 | 93.3
  Would Use Again | 100 | 93.3

8. Secondary Outcome: Percentage of Participants With Anti-Trastuzumab or Anti-Recombinant Human Hyaluronidase (rHuPH20) Antibodies
Description: Participants in Cohort 1 provided blood samples for immunogenicity testing to assess for anti-drug antibodies (ADAs) to trastuzumab or rHuPH20, a component of the SC Herceptin formulation. The percentage of participants who were trastuzumab ADA-positive and the percentage of participants who were rHuPH20 ADA-positive were each reported.
Time Frame: Baseline, pre-dose (0 hours) during Cycle 5 (cycle length of 3 weeks)
Population: Safety Population. Results were planned to be analyzed for only Cohort 1 because the objective of the study was to evaluate immunogenicity within participants who received the SID formulation of Herceptin. The number of participants who provided ADA samples at each timepoint (n) is shown in the table.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: SC (SID) Then IV Herceptin | Cohort 1: IV Then SC (SID) Herceptin
Number analyzed (Participants) | 122 | 122
percentage of participants
  Trastuzumab ADA-Positive, Baseline (n=120,121) | 2.5 | 4.1
  Trastuzumab ADA-Positive, Cycle 5 (n=114,119) | 0 | 3.4
  rHuPH20 ADA-Positive, Baseline (n=120,121) | 5.8 | 7.4
  rHuPH20 ADA-Positive, Cycle 5 (n=115,119) | 2.6 | 7.6

ADVERSE EVENTS:
Time Frame: During treatment from Cycles 1 to 8 (crossover period) and Cycles 9 to 18 (continuation period); cycle length of 3 weeks
Description: Analysis Population Description: Safety Population
Groups:
- Cohort 1: SC (SID) Herceptin (Crossover): Participants received Herceptin on Day 1 of each 3-week cycle for 18 cycles. SC Herceptin was administered via SID as a 600-mg dose during four consecutive cycles of the crossover period. Administration was performed by HCP.
- Cohort 1: IV Herceptin (Crossover); Cohort 2: IV Herceptin (Crossover): Participants received Herceptin on Day 1 of each 3-week cycle for 18 cycles. IV Herceptin was given as a 6-mg/kg dose during four consecutive cycles of the crossover period. If study treatment for Cycle 1 was IV Herceptin, the initial dose was a loading dose of 8 mg/kg (instead of 6 mg/kg) for de novo participants who started Herceptin treatment in the study. Administration was performed by HCP.
- Cohort 1: IV Herceptin (Continuation): Participants received Herceptin on Day 1 of each 3-week cycle for 18 cycles. In the continuation period, participants received IV Herceptin as a 6-mg/kg dose for up to 10 remaining cycles. Administration was performed by HCP.
- Cohort 1: SC (SID) Herceptin (Continuation): Participants received Herceptin on Day 1 of each 3-week cycle for 18 cycles. Those with at least 2 treatment cycles remaining of the 18-cycle treatment course after the crossover period were offered the opportunity to self-administer SC Herceptin via SID as a 600-mg dose under the direction of a trained HCP.
- Cohort 2: SC (Vial) Herceptin (Crossover): Participants received Herceptin on Day 1 of each 3-week cycle for 18 cycles. SC Herceptin was administered via handheld syringe using the vial formulation as a 600-mg dose during four consecutive cycles of the crossover period. Administration was performed by HCP.
- Cohort 2: IV Herceptin (Continuation): Participants received Herceptin on Day 1 of each 3-week cycle for 18 cycles. In the continuation period, participants were planned to receive SC Herceptin via handheld syringe using the vial formulation for up to 10 remaining cycles. However, under protocol deviation a small number of participants received IV Herceptin as a 6-mg/kg dose for this period. Administration was performed by HCP.
- Cohort 2: SC (Vial) Herceptin (Continuation): Participants received Herceptin on Day 1 of each 3-week cycle for 18 cycles. In the continuation period, participants received SC Herceptin via handheld syringe using the vial formulation for up to 10 remaining cycles. Administration was performed by HCP.
Arm/Group | Cohort 1: SC (SID) Herceptin (Crossover) | Cohort 1: IV Herceptin (Crossover) | Cohort 1: IV Herceptin (Continuation) | Cohort 1: SC (SID) Herceptin (Continuation) | Cohort 1 Overall: SC (SID) and IV Herceptin | Cohort 2: SC (Vial) Herceptin (Crossover) | Cohort 2: IV Herceptin (Crossover) | Cohort 2: IV Herceptin (Continuation) | Cohort 2: SC (Vial) Herceptin (Continuation) | Cohort 2 Overall: SC (Vial) and IV Herceptin
Serious Adverse Events (participants affected / at risk) | 4/242 | 2/241 | 6/226 | 1/43 | 12/244 | 0/237 | 2/237 | 0/10 | 5/208 | 7/239
Other Adverse Events (participants affected / at risk) | 81/242 | 55/241 | 46/226 | 7/43 | 130/244 | 107/237 | 76/237 | 6/10 | 61/208 | 154/239
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: SC (SID) Herceptin (Crossover) (N=242) | Cohort 1: IV Herceptin (Crossover) (N=241) | Cohort 1: IV Herceptin (Continuation) (N=226) | Cohort 1: SC (SID) Herceptin (Continuation) (N=43) | Cohort 1 Overall: SC (SID) and IV Herceptin (N=244) | Cohort 2: SC (Vial) Herceptin (Crossover) (N=237) | Cohort 2: IV Herceptin (Crossover) (N=237) | Cohort 2: IV Herceptin (Continuation) (N=10) | Cohort 2: SC (Vial) Herceptin (Continuation) (N=208) | Cohort 2 Overall: SC (Vial) and IV Herceptin (N=239)
Breast abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast reconstruction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Mammoplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Suture related complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: SC (SID) Herceptin (Crossover) (N=242) | Cohort 1: IV Herceptin (Crossover) (N=241) | Cohort 1: IV Herceptin (Continuation) (N=226) | Cohort 1: SC (SID) Herceptin (Continuation) (N=43) | Cohort 1 Overall: SC (SID) and IV Herceptin (N=244) | Cohort 2: SC (Vial) Herceptin (Crossover) (N=237) | Cohort 2: IV Herceptin (Crossover) (N=237) | Cohort 2: IV Herceptin (Continuation) (N=10) | Cohort 2: SC (Vial) Herceptin (Continuation) (N=208) | Cohort 2 Overall: SC (Vial) and IV Herceptin (N=239)
Asthenia (General disorders) | 13 | 10 | 9 | 0 | 30 | 17 | 15 | 0 | 11 | 36
Fatigue (General disorders) | 8 | 10 | 7 | 0 | 23 | 11 | 8 | 1 | 5 | 21
Injection site reaction (General disorders) | 19 | 0 | 0 | 0 | 19 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 13 | 0 | 0 | 0 | 13 | 15 | 0 | 0 | 4 | 17
Injection site pain (General disorders) | 12 | 0 | 0 | 2 | 13 | 20 | 0 | 0 | 6 | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 15 | 12 | 1 | 33 | 15 | 12 | 0 | 10 | 33
Hot flush (Vascular disorders) | 8 | 6 | 3 | 1 | 18 | 14 | 11 | 0 | 5 | 27
Hypertension (Vascular disorders) | 7 | 1 | 5 | 1 | 13 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 14 | 6 | 6 | 1 | 22 | 11 | 8 | 0 | 3 | 17
Headache (Nervous system disorders) | 8 | 6 | 10 | 0 | 21 | 12 | 11 | 0 | 11 | 29
Nasopharyngitis (Infections and infestations) | 5 | 7 | 5 | 1 | 16 | 6 | 3 | 1 | 6 | 13
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 6
Medical device discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 15 | 5 | 0 | 2 | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 4 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 1 | 1 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 4 | 7
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 7 | 0 | 2 | 13
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 2 | 1 | 1 | 11
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 8 | 9 | 0 | 9 | 23
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 15 | 3 | 0 | 6 | 20
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 0 | 6 | 13
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.